CLINICAL TRIAL: NCT04987359
Title: A Randomized Trial of a Multimodal Lifestyle Intervention to Optimize Survivorship After Cancer
Brief Title: A Trial of a Multimodal Lifestyle Intervention to Optimize Survivorship After Cancer
Acronym: Small Steps
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, Justin Brown, Assistant Professor, Pennington Biomedical Research Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PBRC 2021-013
Record Dates: First submitted 2021-07-13; First posted 2021-08-03 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multimodal Lifestyle Program (Experimental): The multimodal lifestyle program will utilize intensive behavioral therapy with structured exercise training and nutritional counseling. The main objective of the structured exercise training is to improve cardiorespiratory fitness.
  Interventions: Behavioral: Multimodal Lifestyle Program
- Waitlist Control (No Intervention): The waitlist control group will be asked to maintain their current exercise and dietary habits for the 10-week study period. Upon providing study endpoint data at week 10, control group participants will be offered a 4-week multimodal lifestyle program that is similar to the intervention group.

INTERVENTIONS:
Behavioral: Multimodal Lifestyle Program — The multimodal lifestyle program will utilize intensive behavioral therapy with structured exercise training and nutritional counseling.
  Arms: Multimodal Lifestyle Program

SUMMARY:
To examine the efficacy of a 10-week multimodal lifestyle program, versus waitlist control, on cardiorespiratory fitness capacity and body weight in survivors of cancer.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent before any trial-related activities
* History of any malignancy
* Completion of cancer-directed therapy (e.g., surgery, chemotherapy, and radiotherapy) prior to enrollment (patients receiving ongoing endocrine or targeted therapy are eligible to participate)
* No evidence of residual or recurrent cancer under active treatment
* Age ≥18 years
* Body mass index (BMI) ≥30 kg/m2 or BMI ≥27 kg/m2 with one or more treated or untreated weight-related coexisting conditions
* Willing to be randomized
* Allow the collection and storage of biospecimens and data for future use

Exclusion Criteria:

* Engaging in ≥3 purposeful exercise sessions per week, on average, over the past 12 weeks
* Significant purposeful weight loss (>11 kg) within the past 12 weeks
* Current use of medications or devices for the purpose of weight loss
* Metabolic or bariatric surgery within the last year
* Cardiovascular, respiratory, or musculoskeletal disease that would prohibit participation in an exercise and weight loss program
* Currently pregnant, breastfeeding, or planning to become pregnant with the next 12 weeks
* Psychiatric disorders or conditions that would preclude participation in the study intervention
* Any other condition which, in the opinion of the investigator, may impede testing of the study hypothesis or make it unsafe to engage in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-08-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in cardiorespiratory fitness capacity (co-primary) | Baseline, Week 10
  Cardiorespiratory fitness (VO2peak) assessed by a symptom-limited cardiopulmonary exercise test.
Change in body weight (co-primary) | Baseline, Week 10
  Bodyweight assessed using a digital scale in a fasting state with an empty bladder, without shoes, and only wearing light clothing.

SECONDARY OUTCOMES:
Change in waist Circumference | Baseline, Week 10
  Measured midway between the lower rib margin and the iliac crest.
Change in fat Mass | Baseline, Week 10
  Measured by dual-energy x-ray absorptiometry
Change in systolic blood pressure | Baseline, Week 10
  Seating, resting for 5 minutes before the measure is taken
Change in diastolic blood pressure | Baseline, Week 10
  Seating, resting for 5 minutes before the measure is taken
Change in medication use | Baseline, Week 10
  Medications related to cholesterol, diabetes, and blood pressure
Change in physical and mental quality-of-life | Baseline, Week 10
  Assessed using the 36-Item Short Form Survey (SF-36)

CONTACTS AND LOCATIONS:
Overall Officials: Justin C Brown, PhD, Principal Investigator — Pennington Biomedical Research Center
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Brown JC, Nauta P, Whitehead D, Dubin BR, Nash R, Blumberg K, Green T, Brown J, Compton SLE, Miletello GP. A randomized trial of a multimodal lifestyle intervention in cancer survivors. Front Oncol. 2025 Oct 2;15:1682244. doi: 10.3389/fonc.2025.1682244. eCollection 2025. PMID 41114371